CLINICAL TRIAL: NCT03890575
Title: Covered Metallic Segmented Airway Stent Modified With 3D Printing for Malignant Stricture Involving Carina and Bronchi Distal to Carina: A Multicenter Study
Brief Title: Airway Segmented Stent Modified With 3D Printing for Malignant Stricture Involving Carina and Distal Bronchi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other); Shanghai Tong Ren Hospital (Other); Ruijin Hospital Luwan Branch (Other)
Responsible Party: Principal Investigator, Zhongmin Wang, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: malignantairwaystent
Record Dates: First submitted 2019-03-19; First posted 2019-03-26 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Stricture; Trachea; Malignant Neoplasm
Keywords: 3D printed; airway stent; carina; distal bronchi
MeSH Terms: conditions — Tracheal Stenosis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Airway Stent for Malignant Stricture (Experimental): Patients with malignant stricture were implanted with covered metallic segmented stent modified with 3D printing.
  Interventions: Procedure: Airway stent implantation

INTERVENTIONS:
Procedure: Airway stent implantation — The airway stents modified with 3D printing were implanted to treat malignant stricture involving carina and bronchi distal to carina.

SUMMARY:
In this study, we used the covered metallic segmented airway stent to treat malignant strictures involving carina and bronchi distal to carina and aimed to determine the feasibility, efficacy and safety of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant stricture involving carina and bronchi distal to carina based on the diagnosis by bronchoscopy or CT.

Exclusion Criteria:

* Severe infection
* Coagulation disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Dyspnea using Hugh-Jones classication as criteria | 3 days
  Hugh-Jones classication: dyspnea scale that includes 5 categories.
Stent patency time | 2 months
  Stent patency time is defined as the time from the stent implantation to stent restenosis or death due to any cause, or censored at date last known alive.
Overall survival | 6 months
  OS is defined as the time from the stent implantation to death due to any cause, or censored at date last known alive.

SECONDARY OUTCOMES:
Number of participants with adverse events that are related to stent implantation | 2 months
  Adverse events as follows: migration of the stent, severe chest pain, hemoptysis, granuloma formation, pneumonia and accumulation of secretion

CONTACTS AND LOCATIONS:
Overall Officials: Zhongmin Wang, MD, Principal Investigator — Ruijin Hospital
Locations (2):
- China (2):
  - Ruijin Hospital Luwan Branch, Shanghai
  - Shanghai Tongren Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No